CLINICAL TRIAL: NCT06442735
Title: Vaginal Delivery Facilitated by Intrapartum Ultrasound During Labor
Brief Title: Clinical Application of Intrapartum Ultrasound
Acronym: IPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ping Li, Clinical Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A2023-264-01
Record Dates: First submitted 2024-05-18; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Abnormal Labor; Complication of Delivery
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapartum ultrasound (Experimental): IPUS group women were performed pelvic examination at admission and every 2 to 4 hours during the first stage of labor and at least hourly during the second stage by intrapartum ultrasound.
  Interventions: Other: intrapartum ultrasound
- Vaginal examination (Active Comparator): VE group women were performed pelvic examination at admission and every 2 to 4 hours during the first stage of labor and at least hourly during the second stage by vaginal examination.
  Interventions: Other: vaginal examination

INTERVENTIONS:
Other: intrapartum ultrasound — In IPUS group, the patient's labor was observed by intrapartum ultrasound.
  Arms: Intrapartum ultrasound
Other: vaginal examination — In VE group, the patient's labor was observed by vaginal examination.
  Arms: Vaginal examination

SUMMARY:
Intrapartum ultrasound monitoring is to be compared with conventional labor monitoring to clarify the accuracy of this technology, and then provide a basis for later related research.

DETAILED DESCRIPTION:
Intrapartum ultrasound monitoring is to be compared with conventional labor monitoring to clarify the accuracy of this technology, and then provide a basis for later related research. All pregnant women intending to have a vaginal delivery were enrolled in the study. After admission, women were randomly assigned to either intrapartum ultrasound (IPUS) or vaginal examination (VE). In IPUS group, the patient was evaluated by ultrasound, including fetal orientation, pelvic and cervical conditions. IPUS and VE were performed every 2 to 4 hours during the first stage of labor and at least hourly during the second stage. The progress of labor, the occurrence of complications and the prediction of the success rate of vaginal delivery were observed. Finally, the investigators compared whether there were any differences in labor and vaginal delivery complications between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in the delivery room for vaginal trial labor

Exclusion Criteria:

* Those who reject ultrasound

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 455 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of the first stage of labor | Day 1
  Medical record about the length of first stage of labor
Duration of the second stage of labor | Day 1
  Medical record about the length of second stage of labor
Number of Participants with fever | Day 3
  physiological parameter about the body temperature when the patient has fever
Number of Participants with the soft birth canal laceration I, II,III, IV | Day 1
  clinical assessment about the soft birth canal laceration after labor, including I(Perineal skin and vaginal entrance mucosa laceration, little bleeding）, II（The lacerated injury has reached the fascia and muscle layer of the perineum, involved the mucous membrane of the posterior wall of the vagina, extended to the groove on both sides of the posterior wall of the vagina and tore upward, the anatomical structure is not easy to identify, and there is more bleeding）,III（The lacerated wound extends deep into the perineum, the external anal sphincter is broken, and the rectal mucosa is intact）, IV（The anus, rectum and vagina are completely penetrated, the rectointestinal cavity is exposed, the histological tissue is seriously damaged）
Number of Participants with postpartum hemorrhage | Day 1
  total postpartum blood loss in 24 hours measured by weighing method

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All data generated or analyzed during this study are available from the Central Contact Person on reasonable request.